CLINICAL TRIAL: NCT02199249
Title: A Prospective Randomized Multi Center Study to Compare Open Reduction, TightRope Fixation (OT) Versus Open Reduction Screw Fixation (OS) of the Tibia - Fibular Syndesmosis.
Brief Title: Open Reduction Syndesmosis Tightrope Versus Screw Fixation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Orthopaedic Trauma Association (Other)
Responsible Party: Principal Investigator, David Sanders, Md, FRCSC, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 105500
Record Dates: First submitted 2014-07-16; First posted 2014-07-24 (Estimated); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Ankle Fractures
Keywords: open anatomic reduction; syndesmosis screw fixation, syndesmosis Tightrope fixation
MeSH Terms: conditions — Ankle Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Open Reduction Tightrope fixation (OT) (Active Comparator): Device: Following fixation of Weber C fibular fracture according to AO standards, the syndesmosis will be stabilized by open reduction followed by use of a single Tightrope (Arthrex-Knotless) device. Open Reduction Tightrope fixation (OT)
  Interventions: Device: Open reduction Tightrope fixation
- Open Reduction screw fixation (OS) (Active Comparator): Device: Following fixation of Weber C fibular fracture according to AO standards, the syndesmosis will be stabilized by open reduction followed by use of two or more syndesmosis screws. Open Reduction screw fixation (OS)
  Interventions: Device: open reduction screw fixation

INTERVENTIONS:
Device: Open reduction Tightrope fixation — Device: Following fixation of Weber C fibular fracture according to AO standards, the syndesmosis will be stabilized by open reduction followed by use of a single Tightrope (Arthrex-Knotless) device. Open Reduction Tightrope fixation (OT)
  Other Names: Athrex tightrope
  Arms: Open Reduction Tightrope fixation (OT)
Device: open reduction screw fixation — Device: Following fixation of Weber C fibular fracture according to AO standards, the syndesmosis will be stabilized by open reduction followed by use of two or more syndesmosis screws. Open Reduction screw fixation (OS)
  Other Names: syndesmosis screw fixation
  Arms: Open Reduction screw fixation (OS)

SUMMARY:
Tibia-fibular syndesmosis injury occurs in a significant proportion of ankle injuries and is assumed to disrupt the syndesmotic ligaments.

The goal of operative treatment is to reduce the ankle mortise to restore normal joint kinematics. Syndesmosis repair can be performed using either open or closed reduction, combined with fixation between the distal tibia and fibula. Closed fixation has demonstrated high rates of non anatomic reductions greater than 40%; therefore, open reduction will be performed in this study. Screw fixation is stable but concerns exist regarding potential excess rigidity.

Recently, flexible fixation techniques combined with anatomic reduction have demonstrated improvements in functional outcomes and reduction quality. Both open reduction and flexible TightRope fixation have considerable support in the literature in cohort studies but have not been compared to open screw fixation in a randomized controlled trial.

In this multi centre randomized study, radiographic, economic and functional outcomes are compared between [open reduction, flexible Tightrope syndesmosis fixation (OT)] and [open reduction screw fixation (OS)] of the syndesmosis.

DETAILED DESCRIPTION:
Tibia-fibular syndesmosis injury occurs in a significant proportion of ankle injuries and is assumed to disrupt the syndesmotic ligaments. The goal of operative treatment is to reduce the ankle mortise to restore normal joint kinematics. Syndesmosis repair can be performed using either open or closed reduction, combined with fixation between the distal tibia and fibula. Closed fixation has demonstrated high rates of non anatomic reductions greater than 40%; therefore, open reduction will be performed in this study. Screw fixation is stable but concerns exist regarding potential excess rigidity.

Recently, flexible fixation techniques combined with anatomic reduction have demonstrated improvements in functional outcomes and reduction quality. Both open reduction and flexible TightRope fixation have considerable support in the literature in cohort studies but have not been compared to open screw fixation in a randomized controlled trial.

This study is a multi centre randomized controlled trial comparing clinical, economic and functional outcomes between open reduction, flexible Tightrope syndesmosis fixation (OT) to open reduction rigid screw fixation (OS) for syndesmotic injuries in high ankle fractures, involving the fibula 1 cm above the level of the syndesmosis (Weber C (OTA 44.C1, 44.C2, 44C3)).

We anticipate recruiting 72 patients (36 in each arm) from up to 20 clinical sites across North America. Post operative follow up will occur at 2 and 6 weeks, 3, 6, and 12 months. At each follow up, radiographic and functional outcomes will be assessed as well as documentation of costs associated with treatment and rehabilitation.

The research questions that this study will answer include the following:

1. Does open reduction and repair with TightRope syndesmosis fixation (OT) provide better reduction compared to open reduction and syndesmosis screw fixation (OS)?
2. Which surgical technique provides better functional outcomes?
3. Are complications and costs associated with repair comparable between surgical techniques?

The null hypothesis is that there will be no difference between the treatment groups in terms of reduction and functional testing.

The scientific aims of this study are to compare:

1. anatomic (open) reduction between the two groups using CT scan and plain radiographs.
2. post-operative pain and functional performance in each group.
3. rates of complications and costs for each method of fixation.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18yrs with a diagnosis of a closed Weber C ankle (OTA 44.C1, 44.C2, 44.C3) fracture.
2. Randomization and treatment of syndesmosis injury within 14 days of the date of injury.
3. Demonstrates lateral subluxation of talus on x-ray or stress views. Talar shift > 1mm or medial clear space widening ≥ 5mm (unstable)
4. No history of previous severe ankle injury, pathologic fracture, ligamentous laxity, no prior diagnosis or current treatment of osteoporosis or metabolic bone disease.
5. No concurrent injury that is deemed by the treating surgeon to delay or alter the rehabilitation protocol for the ankle injury.
6. No neuromuscular or sensory deficiency.
7. Able to understand and complete assessments
8. Provision of Informed Consent

Exclusion Criteria

1. Age < 18 years
2. Open fracture or pathological fracture.
3. Talar shift < 1mm or medial clear space widening < 5mm (stable)
4. Prior diagnosis or current treatment for osteoporosis or metabolic bone disease.
5. Concurrent injury that is deemed by the treating surgeon to delay or alter the rehabilitation protocol for the ankle injury.
6. Prior diagnosis or treatment for neuromuscular disease or sensory deficiency (i.e. diabetic neuropathy).
7. Likely problems, in the judgment of the investigator, with maintaining follow-up (i.e. patients with no fixed address, patients incapable of providing informed consent, prisoners etc.).
8. Patients who are currently pregnant or planning to become pregnant during the study duration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
anatomic reduction between the two groups using CT scan and plain radiographs. | 3 months
  anatomic reduction between the two groups using CT scan and plain radiographs

SECONDARY OUTCOMES:
post-operative pain | 6 weeks, 3, 6, 12 months
  evaluated by means of patient completed visual analogue scale and questionnaires
functional performance | 6 weeks, 3,6 12 months
  patients will complete validated self administered functional outcome, pain and quality of life questionnaires at the time of study enrolment and at 6 weeks, 3, 6 and 12 months following enrolment. Questionnaires will include a generic health status measurement instrument (EQ-5D) and a disease specific outcome measure (Foot and Ankle Disability Index (FADI)). The EQ5D is widely used to describe the extent to which patients are having a problem in each of 5 dimensions of health (mobility, ability to self care, usual activities, pain, and anxiety/depression). The FADI is designed to assess functional limitations related to foot and ankle conditions. It captures activities of daily living and more difficult tasks essential to sport activity (FADI Sport).
  In addition, the AAOS Hindfoot Score will be completed by the surgeon. This score assesses pain, function, alignment, stability and motion. Patients will be asked if they have returned to work with modified duties etc.

CONTACTS AND LOCATIONS:
Overall Officials: David Sanders, MD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

REFERENCES:
- [Derived] Wong MT, Wiens C, LaMothe J, Edwards WB, Schneider PS. In Vivo Syndesmotic Motion After Rigid and Flexible Fixation Using 4-Dimensional Computerized Tomography. J Orthop Trauma. 2022 May 1;36(5):257-264. doi: 10.1097/BOT.0000000000002267. PMID 35594514